CLINICAL TRIAL: NCT01026324
Title: A Phase 1/2 Study of SCH727965 in Patients With Malignant Melanoma
Brief Title: Dinaciclib in Treating Patients With Stage III-IV Melanoma
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2013-00522; NCI-2013-00522 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 09-152 (Other: Dana-Farber Cancer Institute); 8296 (Other: CTEP); U01CA062490 (NIH); P30CA006516 (NIH)
Record Dates: First submitted 2009-12-03; First posted 2009-12-04 (Estimated); Results first posted 2016-08-03 (Estimated); Last update posted 2017-04-04 (Actual); Status verified 2017-03

CONDITIONS: Stage IIIB Melanoma; Stage IIIC Melanoma; Stage IV Melanoma
MeSH Terms: conditions — Melanoma | interventions — dinaciclib

ARMS (1):
- Treatment (dinaciclib) (Experimental): Patients receive dinaciclib IV over 4 hours on day 1. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.
  Interventions: Drug: dinaciclib; Other: pharmacological study; Other: laboratory biomarker analysis

INTERVENTIONS:
Drug: dinaciclib — Given IV
  Other Names: CDK inhibitor SCH 727965; cyclin-dependent kinase inhibitor SCH 727965; SCH 727965
Other: pharmacological study — Correlative studies
  Other Names: pharmacological studies
Other: laboratory biomarker analysis — Correlative studies

SUMMARY:
This is a phase I/II trial is studying the side effects and best dose of dinaciclib and to see how well it works in treating patients with advanced melanoma. Dinaciclib may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the recommended phase 2 dose of SCH727965 administered as a 4-hour infusion every other week in patients with advanced malignant melanoma. (Phase I) II. To determine the 1-year overall survival of patients with malignant melanoma treated with SCH727965 at the dose and schedule derived in the phase 1 part of the study. (Phase II)

SECONDARY OBJECTIVES:

I. To characterize the safety profile and toxicities of SCH727965 administered as a 4-hour infusion every other week.

II. To determine the pharmacokinetics of SCH727965 administered as a 4-hour infusion every other week.

III. To determine the proportion of patients with malignant melanoma who are alive without progression of disease 6 months after beginning treatment with SCH727965 at the dose and schedule derived in the phase 1 part of the study.

IV. To determine the objective response rate to SCH727965 of patients with malignant melanoma enrolled to part 2 of the study.

V. To document cdk2, combined cdk2/1 and cdk9 inhibition in surrogate tissues and tumor.

VI. To correlate the degree of change of pharmacodynamic parameters in post-treatment compared to pre-treatment samples with clinical outcome.

VII. To correlate the degree of change of parameters defining cdk2, cdk2/1 and cdk9 inhibition with pharmacokinetic parameters.

VIII. To correlate pre-treatment cdk2 levels with the degree of change of parameters measuring cdk2 inhibition.

IX. To correlate pre-treatment cdk2 levels with clinical outcome. X. To correlate tumor p53 status with clinical outcome.

OUTLINE: This is a phase I dose-escalation study followed by a phase II study.

Patients receive dinaciclib IV over 4 hours on day 1. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically confirmed, unresectable stage III or stage IV malignant melanoma
* ECOG performance status =< 1
* Absolute neutrophil count >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Total bilirubin within normal institutional limits
* AST(SGOT)/ALT(SGPT =< 1.5 x institutional upper limit of normal
* Creatinine =< 1.5 mg/dl OR
* Creatinine clearance >= 50 mL/min for patients with creatinine levels above institutional normal
* Women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation; should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately
* Eligible patients must agree to pre- and post-treatment biopsies of normal skin; in the phase 1 part of the study, patients with cutaneous disease or accessible lymph nodes must also agree to pre- and post-treatment tumor biopsies; in the phase 2 part of the study, tumor biopsies are required of the first 20 patients enrolled who have cutaneous disease or accessible lymph nodes
* Patients enrolled to the Phase 2 portion of the study must have measurable disease by RECIST criteria
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with active CNS metastases are excluded; patients with a history of CNS metastases that have been treated must be stable for 4 weeks after completion of treatment, with image documentation required; patients must not be taking enzyme-inducing anticonvulsants and must be either off steroids or be receiving a stable dose of steroids
* Uncontrolled intercurrent illness including, but not limited to ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with SCH727965
* HIV-positive patients on combination antiretroviral therapy are ineligible because of the potential for pharmacokinetic interactions with SCH727965; in addition, these patients are at increased risk of lethal infections when treated with marrow-suppressive therapy; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Patients with other currently active malignancies are excluded, except those with an in-situ cancer or basal or squamous cell carcinoma of the skin
* In the phase 2 part of the study, patients who have received prior investigational treatment with a cdk inhibitor are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Frank Hodi, Principal Investigator — Dana-Farber Cancer Institute
Locations (1):
- Dana-Farber Cancer Institute, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were screened and enrolled at one site in the US, Dana Farber Cancer Institute.
Groups:
- Treatment (Dinaciclib) Dose Level 1: Patients receive dinaciclib at Dose Level 1 (10 mg/m2 IV) over 4 hours on day 1. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.
  dinaciclib: Given IV
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Treatment (Dinaciclib) Dose Level 2: Patients receive dinaciclib at Dose Level 2 (20 mg/m2 IV) over 4 hours on day 1. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.
  dinaciclib: Given IV
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
- Treatment (Dinaciclib) Dose Level 3: Patients receive dinaciclib at Dose Level 3(30 mg/m2 IV) over 4 hours on day 1. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.
  dinaciclib: Given IV
  pharmacological study: Correlative studies
  laboratory biomarker analysis: Correlative studies
Period: Treatment Allocation
Arm/Group | Treatment (Dinaciclib) Dose Level 1 | Treatment (Dinaciclib) Dose Level 2 | Treatment (Dinaciclib) Dose Level 3
Started | 5 | 3 | 4
Discontinued Intervention (Toxicity) | 1 | 0 | 0
Discontinuted Intervention (Progression) | 3 | 3 | 4
Discontinued Intervention (Withdrew) | 1 | 0 | 0
Completed | 5 | 3 | 4
Not Completed | 0 | 0 | 0
Period: Follow up/Survival
Arm/Group | Treatment (Dinaciclib) Dose Level 1 | Treatment (Dinaciclib) Dose Level 2 | Treatment (Dinaciclib) Dose Level 3
Started | 5 | 3 | 4
Follow up Discontinuation (Death) | 4 | 3 | 4
Completed | 4 | 3 | 4
Not Completed | 1 | 0 | 0
Not completed — Withdrawal by Subject | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Treatment (Dinaciclib) Dose Level 3: Patients receive dinaciclib at Dose Level 3 (30 mg/m2 IV) over 4 hours on day 1. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.
  dinaciclib: Given IV pharmacological study: Correlative studies laboratory biomarker analysis: Correlative studies
- Total: Total of all reporting groups
Arm/Group | Treatment (Dinaciclib) Dose Level 1 | Treatment (Dinaciclib) Dose Level 2 | Treatment (Dinaciclib) Dose Level 3 | Total
Number analyzed (Participants) | 5 | 3 | 4 | 12
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 4 | 2 | 4 | 10
  >=65 years | 1 | 1 | 0 | 2
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 1 | 5
  Male | 3 | 1 | 3 | 7

OUTCOME MEASURES:

1. Primary Outcome: Recommended Phase-2 Dose of SCH727965
Description: Due to difficult accrual to the trial, enrollment was ended early without determination of an MTD.
Time Frame: 14 days
Population: Due to difficult accrual to the trial, enrollment was ended early without determination of an MTD.
Arm/Group | Treatment (Dinaciclib)
Number analyzed (Participants) | 0

2. Primary Outcome: Percentage of Patients Alive (Phase II)
Description: Due to difficult accrual to the trial, enrollment was ended early without entering into Phase II
Time Frame: Up to 1 year
Population: Due to difficult accrual to the trial, enrollment was ended early without entering into Phase II
Arm/Group | Treatment (Dinaciclib)
Number analyzed (Participants) | 0

3. Secondary Outcome: Progression-free Survival
Time Frame: Up to 6 months
Measure: Number; unit: participants
Groups:
- Treatment (Dinaciclib) Dose Level 1: Patients receive dinaciclib at Dose Level 1 (10 mg/m2 IV) over 4 hours on day 1. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.
  dinaciclib: Given IV
- Treatment (Dinaciclib) Dose Level 2: Patients receive dinaciclib at Dose Level 2 (20 mg/m2 IV) over 4 hours on day 1. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.
  dinaciclib: Given IV
- Treatment (Dinaciclib) Dose Level 3: Patients receive dinaciclib at Dose Level 3 (30 mg/m2 IV) over 4 hours on day 1. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.
  dinaciclib: Given IV
Arm/Group | Treatment (Dinaciclib) Dose Level 1 | Treatment (Dinaciclib) Dose Level 2 | Treatment (Dinaciclib) Dose Level 3
Number analyzed (Participants) | 5 | 3 | 4
participants
  Stable Disease | 2 | 0 | 0
  Progressive Disease | 1 | 3 | 4
  Unevaluable | 2 | 0 | 0

ADVERSE EVENTS:
Groups:
- Dose Level 1 - Treatment (Dinaciclib): Patients receive dinaciclib IV over 4 hours on Day 1. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.
  Dose: 10 MG/M2
  Dinaciclib: Given IV
  Pharmacological study: Correlative studies
  Laboratory biomarker analysis: Correlative studies
- Dose Level 2 - Treatment (Dinaciclib): Patients receive dinaciclib IV over 4 hours on Day 1. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.
  Dose: 20 MG/M2
  Dinaciclib: Given IV
  Pharmacological study: Correlative studies
  Laboratory biomarker analysis: Correlative studies
- Dose Level 3 - Treatment (Dinaciclib): Patients receive dinaciclib IV over 4 hours on Day 1. Courses repeat every 14 days in the absence of disease progression and unacceptable toxicity.
  Dose: 30 MG/M2
  Dinaciclib: Given IV
  Pharmacological study: Correlative studies
  Laboratory biomarker analysis: Correlative studies
Arm/Group | Dose Level 1 - Treatment (Dinaciclib) | Dose Level 2 - Treatment (Dinaciclib) | Dose Level 3 - Treatment (Dinaciclib)
All-Cause Mortality (participants affected / at risk) | 5/5 | 3/3 | 4/4
Serious Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 4/4
Other Adverse Events (participants affected / at risk) | 5/5 | 3/3 | 4/4
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 - Treatment (Dinaciclib) (N=5) | Dose Level 2 - Treatment (Dinaciclib) (N=3) | Dose Level 3 - Treatment (Dinaciclib) (N=4)
Leukocytes (Blood and lymphatic system disorders) | 1 | 1 | 3
Neutrophils (Blood and lymphatic system disorders) | 1 | 3 | 4
Lymphopenia (Blood and lymphatic system disorders) | 0 | 3 | 2
Dehydration (Gastrointestinal disorders) | 0 | 1 | 0
Hyperuricemia (Metabolism and nutrition disorders) | 0 | 1 | 1
Hyponatremia (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypophosphatemia (Metabolism and nutrition disorders) | 1 | 1 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Syncope (Nervous system disorders) | 0 | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Dose Level 1 - Treatment (Dinaciclib) (N=5) | Dose Level 2 - Treatment (Dinaciclib) (N=3) | Dose Level 3 - Treatment (Dinaciclib) (N=4)
Hemoglobin (Blood and lymphatic system disorders) | 2 | 1 | 1
Leukocytes (Blood and lymphatic system disorders) | 2 | 3 | 4
Lymphopenia (Blood and lymphatic system disorders) | 2 | 3 | 2
Neutrophils (Blood and lymphatic system disorders) | 1 | 3 | 4
Hypertension (Cardiac disorders) | 1 | 0 | 0
Hypotension (Cardiac disorders) | 0 | 1 | 0
Fatigue (General disorders) | 3 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 2 | 0 | 1
Anorexia (Gastrointestinal disorders) | 0 | 1 | 0
Dehydration (Gastrointestinal disorders) | 0 | 1 | 1
Diarrhea (Gastrointestinal disorders) | 0 | 2 | 3
Nausea (Gastrointestinal disorders) | 1 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 2 | 2
Edema limb (Blood and lymphatic system disorders) | 1 | 0 | 0
ALT- SGPT (Hepatobiliary disorders) | 2 | 1 | 1
AST- SGOT (Hepatobiliary disorders) | 3 | 2 | 1
Alkaline phosphatase (Hepatobiliary disorders) | 1 | 0 | 0
Bicarbonate (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Hyperglycemia (General disorders) | 3 | 0 | 1
Hyperkalemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hyperuricemia (Renal and urinary disorders) | 2 | 2 | 1
Hypoalbuminemia (Blood and lymphatic system disorders) | 2 | 1 | 0
Hypocalcemia (Blood and lymphatic system disorders) | 2 | 2 | 2
Hypoglycemia (General disorders) | 1 | 0 | 0
Hypokalemia (Blood and lymphatic system disorders) | 3 | 0 | 1
Hypomagnesemia (Blood and lymphatic system disorders) | 1 | 1 | 2
Hyponatremia (Blood and lymphatic system disorders) | 2 | 0 | 0
Hypophosphatemia (Blood and lymphatic system disorders) | 2 | 3 | 1
Syncope (Nervous system disorders) | 0 | 1 | 0
Back-pain (General disorders) | 1 | 0 | 0
Chest wall-pain (General disorders) | 1 | 0 | 0
Head/headache (General disorders) | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less